CLINICAL TRIAL: NCT04598776
Title: Post Market Clinical Follow up Study of CeraRoot Ceramic Implants One-piece: 3 Years Follow up
Brief Title: PMCF Study of CeraRoot Ceramic Implants One-piece: 3 Years Follow up
Status: Completed | Type: Observational
Sponsor: CeraRoot SL (Industry)
Responsible Party: Sponsor
Other Study IDs: 200806
Record Dates: First submitted 2020-09-13; First posted 2020-10-22 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Tooth Loss; Ceramic Implant
Keywords: zirconia implant; zirconium oxide implant; dental implant; ceramic implant; CeraRoot; one-piece; monotype
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective is to evaluate the success / failure rate of CeraRoot ceramic implants (one piece) during three year follow up.

DETAILED DESCRIPTION:
Traditionally the material of choice for dental implants has been titanium. The success of such material has been unquestionable for the last decades. However a number of issues arise lately regarding the biocompatibility or cytotoxicity or allergies regarding the degradation or oxidation particles within the bone or gum. Esthetics has been a concern as well specially in patients with thin biotype where the metal may produce a grayish look of the mucosa. For this reason the dental community and patients have raised much interest in ceramic dental implants as a tooth colored and metal free alternative for dental implants.

Since 2006 CeraRoot ceramic implants have been available in the market.

The reason for designing this PMCF is to evaluate the long term success of CeraRoot ceramic implants

To achieve those objectives an observational study of patients that have received such implant is designed, using marginal bone loss as a primary response variable. It is estimated that a sample size 200 patients over the 3 year period is needed to achieve relevant data.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have received the studied ceramic implant after 27 August 2020.
* Patients of CeraRoot Clinic (Barcelona)
* Age >18
* Single or multiple missing or hopeless teeth

Exclusion Criteria:

* Smokers.
* The patient is taking medications or having treatments which have an effect on healing in general (e.g. steroids, large doses of anti-inflammatory drugs).
* Untreated periodontal conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that needed a tooth replacement that fulfilled the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP OLIVA-OCHOA, MSC, Principal Investigator — CeraRoot SL
Locations (1):
- CeraRoot CLINIC, Les Franqueses del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gahlert M, Roehling S, Sprecher CM, Kniha H, Milz S, Bormann K. In vivo performance of zirconia and titanium implants: a histomorphometric study in mini pig maxillae. Clin Oral Implants Res. 2012 Mar;23(3):281-6. doi: 10.1111/j.1600-0501.2011.02157.x. Epub 2011 Aug 2. PMID 21806681
- [Background] Kohal RJ, Knauf M, Larsson B, Sahlin H, Butz F. One-piece zirconia oral implants: one-year results from a prospective cohort study. 1. Single tooth replacement. J Clin Periodontol. 2012 Jun;39(6):590-7. doi: 10.1111/j.1600-051X.2012.01876.x. Epub 2012 Apr 23. PMID 22519944
- [Background] Payer M, Arnetzl V, Kirmeier R, Koller M, Arnetzl G, Jakse N. Immediate provisional restoration of single-piece zirconia implants: a prospective case series - results after 24 months of clinical function. Clin Oral Implants Res. 2013 May;24(5):569-75. doi: 10.1111/j.1600-0501.2012.02425.x. Epub 2012 Feb 15. PMID 22335358
- [Background] Gahlert M, Burtscher D, Pfundstein G, Grunert I, Kniha H, Roehling S. Dental zirconia implants up to three years in function: a retrospective clinical study and evaluation of prosthetic restorations and failures. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):896-904. doi: 10.11607/jomi.2211. PMID 23748325
- [Background] Siddiqi A, Kieser JA, De Silva RK, Thomson WM, Duncan WJ. Soft and Hard Tissue Response to Zirconia versus Titanium One-Piece Implants Placed in Alveolar and Palatal Sites: A Randomized Control Trial. Clin Implant Dent Relat Res. 2015 Jun;17(3):483-96. doi: 10.1111/cid.12159. Epub 2013 Sep 23. PMID 24112624
- [Background] Hashim D, Cionca N, Courvoisier DS, Mombelli A. A systematic review of the clinical survival of zirconia implants. Clin Oral Investig. 2016 Sep;20(7):1403-17. doi: 10.1007/s00784-016-1853-9. Epub 2016 May 24. PMID 27217032
- [Background] Oliva J, Oliva X, Oliva JD. Five-year success rate of 831 consecutively placed Zirconia dental implants in humans: a comparison of three different rough surfaces. Int J Oral Maxillofac Implants. 2010 Mar-Apr;25(2):336-44. PMID 20369093
- [Background] Oliva J, Oliva X. 15-Year Post-Market Clinical Follow-up Study of 1,828 Ceramic (Zirconia) Implants in Humans. Int J Oral Maxillofac Implants. 2023 Mar-Apr;38(2):357-366. doi: 10.11607/jomi.10000. PMID 37083912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were included if received a CeraRoot implant between August 27th 2020 and December 4th 2023, provided the inclusion criteria were met.
Pre-assignment Details: 98 patients with a total of 175 implants met the inclusion criteria.
Units Other Than Participants: implants
Groups:
- CeraRoot Ceramic Implants: patients that received CeraRoot ceramic implants.
Period: Overall Study
Arm/Group | CeraRoot Ceramic Implants
Started | 98; 175 implants
Completed | 89; 162 implants
Not Completed | 9; 13 implants
Not completed — Protocol Violation | 5
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: Participants received CeraRoot ceramic implant one-piece.
Units Other Than Participants: implants
Groups:
- CeraRoot Implant: CeraRoot ceramic dental implant one-piece
Arm/Group | CeraRoot Implant
Number analyzed (Participants) | 98
Number analyzed (implants) | 175
Age, Customized [Count of Participants; unit: Participants]
  Age <21 | 2
  21-40 | 14
  41-60 | 54
  61-80 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Implants That Survived
Description: Implant without pain, without mobility and in function.
Time Frame: Baseline to 3 years
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Groups:
- CeraRoot Implants: CeraRoot ceramic implants (one-piece)
Arm/Group | CeraRoot Implants
Number analyzed (Participants) | 89
Number analyzed (implants) | 162
implants
  SUCCESS | 157
  FAILURE | 5

2. Secondary Outcome: Number of Implants With Surgical Complications (SC)
Description: Any complications, as bleeding, infection, no primary stability, early loss.... that may appear will be collected
Time Frame: Baseline to 7 days
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Groups:
- CeraRoot Implants: CeraRoot ceramic implants one-piece
Arm/Group | CeraRoot Implants
Number analyzed (Participants) | 89
Number analyzed (implants) | 162
implants | 0

3. Secondary Outcome: Number of Implants With Before Loading Implants Complications (BLIC)
Description: Any complications before the prosthesis is delivered (implant mobility, implant infection, implant loss...) will be collected
Time Frame: 7 days post operative to delivery of prosthesis
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | CeraRoot Implants
Number analyzed (Participants) | 89
Number analyzed (implants) | 162
implants | 0

4. Secondary Outcome: Number of Implants With After Loading Implants Complications (ALIC)
Description: Any complications after the prosthesis is delivered (implant loss, bone loss, implant mobility...) that may appear will be recorded.
Time Frame: From delivery of prosthesis to two years later.
Population: Patients that received CeraRoot implants and were not excluded from the study.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | CeraRoot Implants
Number analyzed (Participants) | 89
Number analyzed (implants) | 162
implants
  Occlusal premature contact | 1
  Premature Loading | 2
  Aseptic Losening | 1
  Sinus Infection | 1

5. Secondary Outcome: Number of Units With Prosthetic Complications (PC)
Description: Any difficulty during the confection of the crown, complications as decementation, chipping, etc... will be registered.
Time Frame: Baseline to 3 years
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | CeraRoot Implants
Number analyzed (Participants) | 89
Number analyzed (implants) | 162
implants | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: FDA protocols for adverse event reporting are considered in this clinical trial in case of need for notification.
Arm/Group | CeraRoot Implants
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-07-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT04598776/Prot_000.pdf